CLINICAL TRIAL: NCT03112642
Title: Does the Use of a Nerve Stimulator Improve the Outcome of Ultrasound-Guided Supraclavicular Block (Anesthesia) for Upper Extremity Surgery?
Brief Title: Nerve Stimulator for Patients With Upper Extremity Disease, Vascular or Orthopedic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: covid pandemic limited participation
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, William Grubb, M.D., Principal Investigator, Associate Professor of Anesthesiology, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0220110040
Record Dates: First submitted 2014-09-03; First posted 2017-04-13 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Other Biomechanical Lesions of Upper Extremity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Group (Active Comparator): In the Standard Group, in the absence of paresthesia and after negative aspiration, the 40 ml of local anesthetic block [0.35% marcaine] will be administered into the brachial plexus of the upper limb being operated on, at the supraclavicular level.
  Interventions: Procedure: Local anesthetic block [0.35% marcaine]
- Test Group (Experimental): In this group, the ultrasound guided local anesthetic block into the brachial plexus at the supraclavicular level of the upper limb being operated on will be supplemented by use of a blockade monitor (Nerve stimulator device) to direct final placement of the needle for the nerve block.
  Only this group of the patients will receive this intervention with sufficient detail so that it can be distinguished from the Test Group
  Interventions: Procedure: Local anesthetic block [0.35% marcaine]; Device: Braun DIG-R-C Stimuplex Blockade Monitor System

INTERVENTIONS:
Procedure: Local anesthetic block [0.35% marcaine] — In the absence of paresthesia and after negative aspiration, the 40 ml of local anesthetic block [0.35% marcaine] will be administered.
  Other Names: 40 ml of local anesthetic block [0.35% marcaine]
Device: Braun DIG-R-C Stimuplex Blockade Monitor System — The blockade system will be initially set at 1 milliamp. As the proximity of the tip of the needle to the components of the brachial plexus becomes evident by ultrasound approximation and the stimulation pattern of the hand and wrist, the output of the system will be reduced to .3-.5 milliamps. With use of the Braun DIG-R-C Stimuplex Blockade Monitor System.
  Arms: Test Group

SUMMARY:
To help determine if there is improved pain relief when a device that makes an arm muscle move (nerve stimulator) is used to place a needle in the area above the collarbone to prevent feeling of pain (anesthesia) of the upper arm.

DETAILED DESCRIPTION:
The Investigators will use the assessment of onset of motor and sensory block Q 5 minutes to distinguish the difference between blocks performed with ultrasound guidance with or without a nerve blockade monitor.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and females 21 through 89
* Agree to study participation and signed the informed consent
* Scheduled for upper extremity surgery with ultrasound guided supraclavicular block -

Exclusion Criteria:

* Children
* Pregnant Women
* Persons with allergies to local anesthetics
* Persons with infections at or near site of needle insertion
* Patients with severe disturbance of cardiac rhythm and heart block
* Patients with severe respiratory compromise
* Patients requiring bilateral upper extremity anesthesia
* Patients with coagulopathy or medical anticoagulation
* Patients with traumatic nerve injury to neck or upper extremity
* Patients with preexisting neurological deficits in the distribution of the block
* Patients with previous surgery to the neck that may distort brachial plexus anatomy

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-11; Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Grubb, DDS, MD, Principal Investigator — Robert Wood Johnson University Hospital
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Group: In this group, the ultrasound guided local anesthetic block into the brachial plexus at the supraclavicular level of the upper limb being operated on will be supplemented by use of a blockade monitor (Nerve stimulator device) to direct final placement of the needle for the nerve block.
  Only this group of the patients will receive this intervention with sufficient detail so that it can be distinguished from the Test Group
  Local anesthetic block [0.35% marcaine]: In the absence of paresthesia and after negative aspiration, the 40 ml of local anesthetic block [0.35% marcaine] will be administered.
  Braun DIG-R-C Stimuplex Blockade Monitor System: The blockade system will be initially set at 1 milliamp. As the proximity of the tip of the needle to the components of the brachial plexus becomes evident by ultrasound approximation and the stimulation pattern of the hand and wrist, the output of the system will be reduced to .3-.5 milliamps. With use of the Braun DIG-R-C Stimuplex Blockade Monitor System.
Period: Overall Study
Arm/Group | Standard Group | Test Group
Started | 6 | 2
Completed | 6 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Group | Test Group | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (12.86) | 61.5 (1.5) | 66.6 (11.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 6 | 1 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Dermatomes With Complete Motor Block of the Upper Extremities at 30 Minutes
Description: dermatomes (with full motor block) will be the outcome measure The investigators will be assessing changes between muscle strength in the myotomal distribution of the upper limb corresponding to the dermatome region of the brachial plexus following supraclavicular block, using the MRC power scale (medical research council scale, 0-5), with strength values obtained at time zero (initiation of the block), and to compared to subsequent measurements in 5 minute intervals until the final measurement at 30 minutes following the block.
Time Frame: 30 minutes post block
Population: Dermatomes
Measure: Count of Units; unit: dermatomes
Units Other Than Participants: dermatomes
Arm/Group | Standard Group | Test Group
Number analyzed (Participants) | 6 | 2
Number analyzed (dermatomes) | 18 | 6
dermatomes | 18 | 6

2. Other Pre Specified Outcome: Dermatomes With Response to Fine Touch at 30 Minutes
Description: The investigators are assessing changes response to fine touch provocation in the dermatomal distribution of the upper limb corresponding to the anesthetized region of the brachial plexus following supraclavicular block, using a sterile non penetrating (blunt tip) needle and recording responses on a binary scale of sensation (can or cannot feel fine touch stimulus), with sensory values obtained at time zero (initiation of the block), and to compared to subsequent measurements in 5 minute intervals until the final measurement at 30 minute following the block.
Time Frame: 30 minutes post block
Population: Dermatomes with a response to fine touch at 30 minutes
Measure: Count of Units; unit: dermatomes
Units Other Than Participants: dermatomes
Arm/Group | Standard Group | Test Group
Number analyzed (Participants) | 6 | 2
Number analyzed (dermatomes) | 18 | 6
dermatomes | 18 | 6

ADVERSE EVENTS:
Time Frame: 1 week
Description: no difference
Arm/Group | Standard Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 0/6 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT03112642/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT03112642/SAP_001.pdf
  • Informed Consent Form (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT03112642/ICF_002.pdf